CLINICAL TRIAL: NCT01262846
Title: Improving Immunogenicity of Influenza Vaccine in HIV Infected Individuals
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UPenn FLU 02
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: HIV Infection
Keywords: HIV; Flu vaccination; HIV infected individuals; Fluzone SD; Fluzone HD
MeSH Terms: conditions — HIV Infections; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone SD (Active Comparator): Fluzone® Standard dose
  Interventions: Biological: Fluzone®
- Fluzone® High dose (Experimental): Fluzone® High dose in a blinded manner as single-0.5mL injection intramuscularly into one of the subject's deltoid muscles.
  Interventions: Biological: Fluzone®

INTERVENTIONS:
Biological: Fluzone® — Fluzone® Standard dose in a blinded manner as single-0.5mL injection intramuscularly into one of the subject's deltoid muscles.
  Arms: Fluzone SD
Biological: Fluzone® — Fluzone® High dose or Standard dose in a blinded manner as single-0.5mL injection intramuscularly into one of the subject's deltoid muscles.
  Arms: Fluzone® High dose

SUMMARY:
The overall goal of this study is to compare the safety and immunogenicity of trivalent Fluzone® High-Dose vaccine vs the regular standard-dose (SD) in HIV infected individuals. Our hypothesis is that Fluzone® HD will be safe and more immunogenic than the currently used vaccine

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of HIV-1 infection as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry or any measurable HIV RNA viral load in the chart. Serum HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
2. > 18 years
3. Able to understand and comply with planned study procedures.
4. Provides written informed consent prior to initiation of any study procedures.
5. Subject should be 1) on stable antiretroviral therapy as outlined in the DHHS treatment guidelines for HIV-1 infected individuals OR 2) not on antiretroviral therapy and not intending to start treatment within the next 30 days.

Exclusion Criteria:

1. Has a known allergy to eggs or other components in the vaccines (these may include, but are not limited to: gelatin, formaldehyde, octoxinol and chicken protein).
2. Has a history, in the opinion of the site investigator, of severe reactions following previous immunization with seasonal TIV.
3. Participation in a novel H1N1 influenza vaccine study in the past two years.
4. Proven history, by RT-PCR, of novel influenza H1N1 infection, or, has a positive influenza diagnostic testing since June 2009 (specificity to H1N1 not required) prior to study entry.
5. Received any other live licensed vaccine within 4 weeks or inactivated licensed vaccine within 1 week prior to study entry.
6. Scheduled administration of any live virus vaccine or inactivated vaccine at or between entry and the Day 21 visit. NOTE: Live or inactivated vaccines expected to be administered between study entry and the Day 21 visit should be excluded to prevent potential interference with immunogenicity responses and confounding safety results.
7. Received a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) within 4 weeks prior to vaccination in this study with the exception of new antiretroviral medications as part of a phase 3 trial.
8. An acute illness and/or an oral temperature greater than or equal to 100.0 degrees F within 24 hours prior to study entry.
9. Use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months of study enrollment, or has immunosuppression as a result of an underlying illness or treatment (other than HIV-1 infection).
10. Active neoplastic disease (excluding non-melanoma skin cancer, and HPV-related cervical dysplasia, CIN grades 1, 2 or 3).
11. Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry. NOTE: Subjects receiving stable physiologic glucocorticoid doses, defined as prednisone ≤10 mg/day, will not be excluded. Subjects receiving corticosteroids for acute therapy for an opportunistic infection such as Pneumocystis jiroveci pneumonia (PCP), or receiving a short course (defined as ≤2 weeks) of pharmacologic glucocorticoid therapy will not be excluded.
12. Received immunoglobulin or other blood products
13. Current diagnosis of uncontrolled major psychiatric disorder.
14. History of Guillain-Barré Syndrome in the subject or subject's family (parents, siblings, half siblings, or children).
15. Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PABLO TEBAS, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Clinical Trials Unit. University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Tebas P, Frank I, Lewis M, Quinn J, Zifchak L, Thomas A, Kenney T, Kappes R, Wagner W, Maffei K, Sullivan K; Center for AIDS Research and Clinical Trials Unit of the University of Pennsylvania. Poor immunogenicity of the H1N1 2009 vaccine in well controlled HIV-infected individuals. AIDS. 2010 Sep 10;24(14):2187-92. doi: 10.1097/QAD.0b013e32833c6d5c. PMID 20616698
- [Result] McKittrick N, Frank I, Jacobson JM, White CJ, Kim D, Kappes R, DiGiorgio C, Kenney T, Boyer J, Tebas P. Improved immunogenicity with high-dose seasonal influenza vaccine in HIV-infected persons: a single-center, parallel, randomized trial. Ann Intern Med. 2013 Jan 1;158(1):19-26. doi: 10.7326/0003-4819-158-1-201301010-00005. PMID 23277897

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluzone SD | Fluzone® High Dose
Started | 95 | 100
Completed | 93 | 97
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone SD | Fluzone® High Dose | Total
Number analyzed (Participants) | 95 | 100 | 195
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [37 to 53] | 44 [35 to 50] | 45 [35 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 36 | 58
  Male | 73 | 64 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 88 | 97 | 185
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 58 | 78 | 136
  White | 36 | 22 | 58
  More than one race | 0 | 00 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity
Description: To compare the immunogenicity of trivalent Fluzone® High-Dose vaccine vs the regular standard-dose (SD) in HIV infected individuals.
Time Frame: Baseline to 21 days
Population: All participants except 5 participants with missing data at day 21
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean antibody titer
Groups:
- SD Recipients: Fluzone Regular Dose
- HD Recipients: Fluzone High Dose
Arm/Group | SD Recipients | HD Recipients
Number analyzed (Participants) | 93 | 97
Geometric Mean antibody titer
  Baseline H1N1 (A/California/07/2009 X-179 A) | 22 [14 to 37] | 25 [15 to 40]
  Week 3 H1N1 (A/California/07/2009 X-179 A) | 344 [229 to 518] | 686 [509 to 926]
  Baseline H3N2 A/Victoria/210/2009 X-187 | 25 [16 to 42] | 26 [16 to 42]
  Week 3 H3N2 A/Victoria/210/2009 X-187 | 324 [227 to 464] | 739 [529 to 1032]
  Baseline B/Brisbane/60/2008 (influenza B) | 17 [11 to 25] | 20 [14 to 28]
  Week 3 B/Brisbane/60/2008 (influenza B) | 64 [46 to 91] | 140 [110 to 178]

ADVERSE EVENTS:
Arm/Group | SD Recipients | HD Recipients
Serious Adverse Events (participants affected / at risk) | 3/95 | 0/100
Other Adverse Events (participants affected / at risk) | 73/95 | 90/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SD Recipients (N=95) | HD Recipients (N=100)
Hospitalization (General disorders) | 3 | 0
Death (General disorders) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SD Recipients (N=95) | HD Recipients (N=100)
Pain (Skin and subcutaneous tissue disorders) | 4 (4) | 15 (15) — Local at injection site
Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Local at injection site
Induration (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) — Local
Tenderness (Skin and subcutaneous tissue disorders) | 10 (10) | 10 (10) — Local
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Chills (General disorders) | 3 (3) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 7 (7)
Headache (General disorders) | 9 (9) | 8 (8)
Lymphadenopathy (Infections and infestations) | 1 (1) | 0 (0)
Malaise (General disorders) | 14 (14) | 13 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (17) | 19 (19)
vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Caution The trial was not powered to determine clinical efficacy or to detect differences in the occurrence of less common adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No